CLINICAL TRIAL: NCT06077760
Title: A Phase 3, Randomized, Double-blind, Placebo- and Active-Comparator-Controlled Clinical Study of Adjuvant V940 (mRNA-4157) Plus Pembrolizumab Versus Adjuvant Placebo Plus Pembrolizumab in Participants With Resected Stage II, IIIA, IIIB (N2) Non-small Cell Lung Cancer (INTerpath-002)
Brief Title: A Study of Intismeran Autogene (V940) Plus Pembrolizumab (MK-3475) Versus Placebo Plus Pembrolizumab in Participants With Non-small Cell Lung Cancer (V940-002)
Acronym: INTerpath-002
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: V940-002; 2023-504923-20-00 (Registry Identifier: EU CT); U1111-1290-3969 (Registry Identifier: UTN); jRCT2061240063 (Registry Identifier: jRCT); PHRR240705-007252 (Registry Identifier: PHRR)
Record Dates: First submitted 2023-10-05; First posted 2023-10-11 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intismeran autogene + Pembrolizumab (Experimental): Participants will receive 1 mg of intismeran autogene via intramuscular (IM) injection once every 3 weeks for 9 doses PLUS 400 mg of pembrolizumab via intravenous (IV) infusion once every 6 weeks for up to 9 doses until disease recurrence or unacceptable toxicity or for a total treatment duration of up to approximately 1 year, whichever is sooner.
  Interventions: Biological: Intismeran autogene; Biological: Pembrolizumab
- Placebo + Pembrolizumab (Active Comparator): Participants will receive intismeran autogene-matched placebo via IM injection once every 3 weeks for 9 doses PLUS 400 mg of pembrolizumab via IV infusion once every 6 weeks for up to 9 doses until disease recurrence or unacceptable toxicity or for a total treatment duration of up to approximately 1 year, whichever is sooner.
  Interventions: Biological: Pembrolizumab; Other: Placebo

INTERVENTIONS:
Biological: Intismeran autogene — IM injection
  Other Names: mRNA-4157; V940
  Arms: Intismeran autogene + Pembrolizumab
Biological: Pembrolizumab — IV infusion
  Other Names: MK-3475; KEYTRUDA®
Other: Placebo — IM injection
  Arms: Placebo + Pembrolizumab

SUMMARY:
The goal of this study is to evaluate intismeran autogene plus pembrolizumab versus placebo plus pembrolizumab for the adjuvant treatment of margin negative, completely resected Stage II, IIIA, IIIB (with nodal involvement [N2]) non-small cell lung cancer (NSCLC). The primary hypothesis is that intismeran autogene plus pembrolizumab is superior to placebo plus pembrolizumab with respect to disease-free survival (DFS) as assessed by the investigator.

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

* Has undergone margin negative, completely resected non-small cell lung cancer (NSCLC), and has pathological Stage II, IIIA, IIIB (N2) squamous or nonsquamous tumor, node, metastasis (TNM) staging per American Joint Committee on Cancer (AJCC) Eighth Edition guidelines.
* Has no evidence of disease before randomization.
* Has received at least one dose of adjuvant treatment with standard of care platinum doublet chemotherapy.
* No more than 24 weeks have elapsed between surgical resection of curative intent and the first dose of pembrolizumab.
* Participants who are hepatitis B surface antigen (HBsAg) positive are eligible if they have received hepatitis B virus (HBV) antiviral therapy for at least 4 weeks and have undetectable HBV viral load prior to randomization.
* Participants with history of hepatitis C virus (HCV) infection are eligible if HCV viral load is undetectable at screening.
* Human immunodeficiency virus (HIV)-infected participants must have well controlled HIV on anti-retroviral therapy (ART).

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* Diagnosis of small cell lung cancer (SCLC) or, for mixed tumors, presence of small cell elements, or has a neuroendocrine tumor with large cell components or a sarcomatoid carcinoma.
* HIV-infected participants with a history of Kaposi's sarcoma and/or Multicentric Castleman's Disease.
* Received prior neoadjuvant therapy for their current NSCLC diagnosis.
* Received or is a candidate to receive radiotherapy for their current NSCLC diagnosis.
* Received prior therapy with an anti-programmed cell death 1 protein (PD-1), anti-PD-ligand 1 (L1), or anti-PD-L2 agent, or with an agent directed to another stimulatory or coinhibitory T-cell receptor.
* Received prior systemic anticancer therapy including investigational agents within 4 weeks before randomization.
* Received a live or live-attenuated vaccine within 30 days before the first dose of study intervention. Administration of killed vaccines are allowed.
* Has received an investigational agent or has used an investigational device within 4 weeks prior to study intervention administration.
* Diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study medication.
* Known additional malignancy that is progressing or has required active treatment within the past 5 years.
* Active autoimmune disease that has required systemic treatment in the past 2 years. Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid) is allowed.
* History of (noninfectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
* Active infection requiring systemic therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 868 (Estimated)
Dates: Start 2023-12-06 (Actual); Primary Completion 2030-06-25 (Estimated); Study Completion 2035-12-21 (Estimated)

PRIMARY OUTCOMES:
Disease- Free Survival (DFS) | Up to ~78 months
  DFS is defined as the time from randomization to any recurrence (local, locoregional, regional or distant), occurrence of new primary NSCLC, as assessed by the investigator, or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to ~12 years
  OS is defined as the time from randomization to death due to any cause.
Distant Metastasis-Free Survival (DMFS) | Up to ~12 years
  DMFS is defined as the time from randomization to the first diagnosis of a distant metastasis as assessed by the investigator, or death due to any cause, whichever occurs first.
Lung Cancer Specific Survival (LCSS) | Up to ~12 years
  LCSS is defined as the time from randomization to death due to lung cancer.
Change from Baseline in the European Organization for Research and Treatment of Cancer (EORTC)-Quality of Life Questionnaire-Core 30 (QLQ-C30) Global Health Status/Quality of Life (Items 29 and 30) Combined Score | Baseline and up to ~12 years
  The EORTC QLQ-C30 is a 30-item questionnaire to assess the overall quality of life of cancer patients. Participant responses to the questions "How would you rate your overall health during the past week?" and "How would you rate your overall quality of life during the past week?" will be scored on a 7-point scale (1= Very poor to 7=Excellent). Using linear transformation, raw scores will be standardized, so that scores range from 0 to 100. Higher scores indicate a better overall health status. The change from baseline in global health status/quality of life (EORTC QLQ-C30 Items 29 and 30) combined score will be presented.
Change from Baseline in the EORTC QLQ-C30 Physical Functioning (Items 1-5) Combined Score on the EORTC QLQ-C30 | Baseline and up to ~12 years
  The EORTC QLQ-C30 is a 30-item questionnaire to assess the overall quality of life of cancer patients. Participant responses to 5 questions about their physical functioning will be scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores will be standardized, so that scores range from 0 to 100. Higher scores indicate a worse level of physical functioning. The change from baseline in physical functioning (EORTC QLQ-C30 Items 1-5) combined score will be presented.
Change from Baseline in the EORTC QLQ-C30 Role Functioning (Items 6 and 7) Combined Score on the EORTC QLQ-C30 | Baseline and up to ~12 years
  The EORTC QLQ-C30 is a 30-item questionnaire to assess the overall quality of life of cancer patients. Participant responses to the questions "Were you limited in doing either your work or other daily activities during the past week?" and " Were you limited in pursuing your hobbies or other leisure time activities during the past week?" will be scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores will be standardized, so that scores range from 0 to 100. Higher scores indicate a worse level of role functioning. The change from baseline in role functioning (EORTC QLQ-C30 Items 6 and 7) combined score will be presented.
Change from Baseline in the EORTC QLQ-C30 Dyspnea (Item 8) Score on the EORTC QLQ-C30 | Baseline and up to ~12 years
  The EORTC QLQ-C30 is a 30-item questionnaire to assess the overall quality of life of cancer patients. Participant responses to the question "Were you short of breath?" will be scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores will be standardized, so that scores range from 0 to 100. Higher scores indicate a worse level of dyspnea. The change from baseline in dyspnea (EORTC QLQ-C30 Item 8) score will be presented.
Change from Baseline in the EORTC QLQ-Lung Cancer Questionnaire (LC24) Coughing (Items 31 and 52) Combined Score on the EORTC QLQ-LC24 | Baseline and up to ~12 years
  The EORTC QLQ-LC24 is a lung cancer specific health-related quality of life questionnaire. Participant responses to questions about coughing will be scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores will be standardized, so that scores range from 0 to 100. A higher score indicates more coughing. The change from baseline in coughing (EORTC QLQ-LC24 Items 31 and 52) combined score will be presented.
Change from Baseline in the EORTC QLQ-LC24 Chest Pain (Item 40) Score on the EORTC QLQ-LC24 | Baseline and up to ~12 years
  The EORTC QLQ-LC24 is a lung cancer specific health-related quality of life questionnaire. Participant responses to the question "Have you had pain in your chest?" will be scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores will be standardized, so that scores range from 0 to 100. A higher score indicates more chest pain. The change from baseline in chest pain (EORTC QLQ-LC24 Item 40) score will be presented.
Number of Participants Who Experience an Adverse Event (AE) | Up to ~15 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Number of Participants Who Discontinue Study Treatment Due to an AE | Up to ~12 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (223):
- United States (65):
  - Alaska Oncology and Hematology ( Site 0039), Anchorage, Alaska
  - The University of Arizona Cancer Center - North Campus ( Site 0071), Tucson, Arizona
  - YUMA REGIONAL MEDICAL CENTER CANCER CENTER ( Site 0020), Yuma, Arizona
  - UCLA Clinical & Translational Research Center (CTRC) ( Site 0059), Los Angeles, California
  - Hoag Memorial Hospital Presbyterian ( Site 4042), Newport Beach, California
  - Hoag Memorial Hospital Presbyterian ( Site 4048), Newport Beach, California
  - St. Joseph Hospital-The Center for Cancer Prevention and Treatment ( Site 0074), Orange, California
  - University of California, Irvine (UCI) Health - UC Irvine Medical Center ( Site 0030), Orange, California
  - UCHealth Memorial Hospital-Heme Onc ( Site 0052), Colorado Springs, Colorado
  - Mayo Clinic Florida ( Site 4043), Jacksonville, Florida
  - Mid Florida Hematology and Oncology Center ( Site 0014), Orange City, Florida
  - AdventHealth Orlando-AdventHealth Medical Group Hematology & Oncology at Orlandoc ( Site 0013), Orlando, Florida
  - Moffitt Cancer Center ( Site 0078), Tampa, Florida
  - Northwest Georgia Oncology Centers, a Service of Wellstar Cobb Hospital ( Site 0012), Marietta, Georgia
  - Southeastern Regional Medical Center ( Site 0098), Newnan, Georgia
  - Beacon Cancer Care ( Site 0044), Post Falls, Idaho
  - Illinois Cancer Care ( Site 7003), Peoria, Illinois
  - University of Iowa-Holden Comprehensive Cancer Center ( Site 0062), Iowa City, Iowa
  - Saint Elizabeth Healthcare ( Site 0092), Edgewood, Kentucky
  - The University of Louisville, James Graham Brown Cancer Center ( Site 0037), Louisville, Kentucky
  - LSU Health Baton Rouge North Clinic ( Site 4040), Baton Rouge, Louisiana
  - Our Lady of the Lake RMC-Clinical Research ( Site 4050), Baton Rouge, Louisiana
  - University of Michigan Clinical Trials Office ( Site 0058), Ann Arbor, Michigan
  - Cancer and Hematology Centers of Western Michigan ( Site 4003), Grand Rapids, Michigan
  - St. Vincent Frontier Cancer Center ( Site 0043), Billings, Montana
  - NHO Revive Research Institute, LLC ( Site 4009), Lincoln, Nebraska
  - Memorial Sloan Kettering - Basking Ridge ( Site 4056), Basking Ridge, New Jersey
  - John Theurer Cancer Center at Hackensack University Medical Center ( Site 0036), Hackensack, New Jersey
  - Memorial Sloan Kettering - Monmouth ( Site 4057), Middletown, New Jersey
  - Memorial Sloan Kettering - Bergen ( Site 4059), Montvale, New Jersey
  - Atlantic Health Morristown Medical Center ( Site 4018), Morristown, New Jersey
  - New York Oncology Hematology, P.C. ( Site 4012), Albany, New York
  - Memorial Sloan-Kettering Cancer Center at Commack ( Site 4055), Commack, New York
  - Memorial Sloan Kettering - Westchester ( Site 4058), Harrison, New York
  - Perlmutter Cancer Center at NYU Langone Hospital - Long Island-Clinical Research Department ( Site 0095), Mineola, New York
  - The Blavatnik Family- Chelsea Medical Center at Mount Sinai ( Site 4053), New York, New York
  - Laura and Isaac Perlmutter Cancer Center ( Site 0010), New York, New York
  - Icahn School of Medicine at Mount Sinai ( Site 0034), New York, New York
  - Columbia University Irving Medical Center-CUIMC Herbert Irving Comprehensive Cancer Center Clinical ( Site 0054), New York, New York
  - Memorial Sloan Kettering Cancer Center ( Site 0029), New York, New York
  - Stony Brook University-Cancer Center ( Site 0072), Stony Brook, New York
  - Montefiore Medical Center- Montefiore Medical Park-Oncology ( Site 0080), The Bronx, New York
  - Memorial Sloan Kettering - Nassau ( Site 4060), Uniondale, New York
  - Novant Health Weisiger Cancer Insititute ( Site 4052), Charlotte, North Carolina
  - Novant Health Oncology Specialists ( Site 4045), Winston-Salem, North Carolina
  - Sanford Fargo Medical Center-Roger Maris Cancer Center ( Site 0063), Fargo, North Dakota
  - Altru Health System ( Site 0040), Grand Forks, North Dakota
  - Summa Health ( Site 4011), Akron, Ohio
  - University of Cincinnati Medical Center-University of Cincinnati Cancer Center ( Site 0028), Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center ( Site 0023), Cleveland, Ohio
  - OSU Brain and Spine Hospital ( Site 0016), Columbus, Ohio
  - Good Samaritan Regional Medical Center-Samaritan Pastega Regional Cancer Center ( Site 0082), Corvallis, Oregon
  - Thomas Jefferson University - Clinical Research Institute ( Site 0006), Philadelphia, Pennsylvania
  - Medical University of South Carolina-Hollings Cancer Center ( Site 0050), Charleston, South Carolina
  - Sanford Cancer Center ( Site 0075), Sioux Falls, South Dakota
  - Thompson Cancer Survival Center ( Site 0097), Knoxville, Tennessee
  - Baptist Cancer Center ( Site 4049), Memphis, Tennessee
  - One Oncology - Tennessee Oncology ( Site 4019), Nashville, Tennessee
  - SCRI Oncology Partners ( Site 7001), Nashville, Tennessee
  - UT Southwestern Medical Center ( Site 0061), Dallas, Texas
  - Inova Schar Cancer Institute ( Site 0003), Fairfax, Virginia
  - Virginia Cancer Specialists (VCS) ( Site 4004), Fairfax, Virginia
  - Swedish Medical Center-Swedish Cancer Institute ( Site 0088), Seattle, Washington
  - Fred Hutchinson Cancer Center ( Site 0002), Seattle, Washington
  - Edwards Comprehensive Cancer Center ( Site 4015), Huntington, West Virginia
- Argentina (6):
  - Clinica Adventista Belgrano-Oncology ( Site 2901), Caba., Buenos Aires
  - Hospital Italiano de Buenos Aires-Clinical Oncology ( Site 2912), Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Instituto Alexander Fleming ( Site 2911), Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Instituto de Investigaciones Clínicas Mar del Plata ( Site 2908), Mar del Plata, Buenos Aires
  - Fundacion Estudios Clinicos-Oncology ( Site 2907), Rosario, Santa Fe Province
  - Sanatorio Parque ( Site 2904), Rosario, Santa Fe Province
- Australia (3):
  - Peter MacCallum Cancer Centre-Parkville Cancer Clinical Trials Unit (PCCTU) ( Site 0203), Melbourne, Victoria
  - St Vincent's Hospital-Oncology Clinical Trials ( Site 0202), Melbourne, Victoria
  - One Clinical Research ( Site 0200), Nedlands, Western Australia
- Belgium (4):
  - Antwerp University Hospital-Thoracic Oncology ( Site 0603), Edegem, Antwerpen
  - Université Catholique de Louvain-Namur - Centre Hospitalier Universitaire Dinant-Godinne - Site Godi ( Site 0602), Yvoir, Namur
  - AZORG Campus Aalst-Moorselbaan ( Site 0604), Aalst, Oost-Vlaanderen
  - VITAZ ( Site 0600), Sint-Niklaas, Oost-Vlaanderen
- Brazil (9):
  - CRIO - CENTRO REGIONAL INTEGRADO DE ONCOLOGIA-Pesquisa Clínica ( Site 3007), Fortaleza, Ceará
  - Liga Norte Riograndense Contra o Câncer ( Site 3001), Natal, Rio Grande do Norte
  - Irmandade da Santa Casa de Misericórdia de Porto Alegre ( Site 3003), Porto Alegre, Rio Grande do Sul
  - Hospital Nossa Senhora da Conceição ( Site 3002), Porto Alegre, Rio Grande do Sul
  - Fundação Pio XII - Hospital de Câncer de Barretos ( Site 3004), Barretos, São Paulo
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto ( Site 3013), São José do Rio Preto, São Paulo
  - Instituto Nacional de Câncer - INCA ( Site 3000), Rio de Janeiro
  - Hospital Samaritano De Sao Paulo ( Site 3006), São Paulo
  - ICESP - INSTITUTO DO CÂNCER DO ESTADO DE SÃO PAULO ( Site 3005), São Paulo
- Canada (5):
  - Cross Cancer Institute ( Site 0105), Edmonton, Alberta
  - William Osler Health System ( Site 0101), Brampton, Ontario
  - Princess Margaret Cancer Centre ( Site 0102), Toronto, Ontario
  - Centre Hospitalier de l'Université de Montréal ( Site 0104), Montreal, Quebec
  - McGill University Health Centre ( Site 0100), Montreal, Quebec
- Chile (5):
  - Orlandi Oncologia-Oncology ( Site 3102), Santiago, Region M. de Santiago
  - FALP-UIDO ( Site 3100), Santiago, Region M. de Santiago
  - Pontificia Universidad Catolica de Chile ( Site 3104), Santiago, Region M. de Santiago
  - Bradfordhill-Clinical Area ( Site 3103), Santiago, Region M. de Santiago
  - ONCOCENTRO APYS ( Site 3105), Viña del Mar, Región de Valparaíso
- Costa Rica (2):
  - CIMCA ( Site 3300), San José, Provincia de San José
  - ICIMED ( Site 3301), San José
- Czechia (4):
  - Masarykuv onkologicky ustav-Klinika komplexni onkologicke pece ( Site 0700), Brno, Brno-mesto
  - Nemocnice AGEL Ostrava - Vitkovice a.s.-Plicni odd ( Site 0702), Ostrava, Ostrava Mesto
  - Fakultni nemocnice Olomouc-Klinika plicnich nemoci a tuberkulozy ( Site 0701), Olomouc
  - Vseobecna fakultni nemocnice v Praze ( Site 0703), Prague
- Denmark (2):
  - Rigshospitalet ( Site 0801), Copenhagen, Capital Region
  - Odense Universitetshospital ( Site 0800), Odense, Region Syddanmark
- Estonia (2):
  - North Estonia Medical Centre Foundation-Chemotherapy ( Site 0901), Tallinn, Harju
  - Tartu University Hospital-Radiotherapy and oncology ( Site 0900), Tartu, Tartu
- Finland (4):
  - Oulun yliopistollinen sairaala-Oncology and Hematology ( Site 1003), Oulu, North Ostrobothnia
  - Tampereen yliopistollinen sairaala-Oncology ( Site 1001), Tampere, Pirkanmaa
  - Vaasan Keskussairaala-Department of Clinical Oncology ( Site 1004), Vaasa, Pohjanmaa
  - Turku University Hospital-The Department of Pulmonary Medicine ( Site 1000), Turku, Southwest Finland
- France (8):
  - Nouvel Hôpital Civil (NHC)-Service de pneumologie ( Site 1100), Strasbourg, Alsace
  - CHU Bordeaux Haut-Leveque ( Site 1106), Pessac, Aquitaine
  - Assistance Publique Hôpitaux de Marseille - Hôpital Nord ( Site 1108), Marseille, Bouches-du-Rhone
  - Centre Hospitalier Universitaire de Caen - Hôpital Côte de Nacre ( Site 1107), Caen, Calvados
  - Hôpital Arnaud de Villeneuve - CHU Montpellier ( Site 1102), Montpellier, Herault
  - Institut de Cancérologie de l'Ouest ( Site 1101), Angers, Maine-et-Loire
  - CHU GABRIEL MONTPIED ( Site 1105), Clermont-Ferrand, Puy-de-Dome
  - Hopitaux Universitaires Paris Centre-Hopital Cochin ( Site 1104), Paris
- Germany (10):
  - Klinikum Esslingen-Klinik für Kardiologie und Pneumologie ( Site 1201), Esslingen am Neckar, Baden-Wurttemberg
  - Asklepios Klinik Gauting GmbH-Oncology ( Site 1209), Gauting, Bavaria
  - Klinikverbund Allgäu gGmbH ( Site 1205), Kempten (Allgäu), Bavaria
  - Universitaetsklinikum Regensburg ( Site 1204), Regensburg, Bavaria
  - Augusta-Kranken-Anstalt ( Site 1213), Bochum, North Rhine-Westphalia
  - Gemeinschaftspraxis für Hämatologie und Onkologie Münster ( Site 1202), Münster, North Rhine-Westphalia
  - Brüderkrankenhaus St. Josef Paderborn-Klinik für Hämatologie und Onkologie ( Site 1214), Paderborn, North Rhine-Westphalia
  - LungenClinic Grosshansdorf-Onkologie ( Site 1203), Großhansdorf, Schleswig-Holstein
  - SRH Wald-Klinikum Gera-Lungenkrebszentrum ( Site 1200), Gera, Thuringia
  - Helios Klinikum Emil von Behring Berlin-Zehlendorf-Lungenklinik Heckeshorn ( Site 1208), Berlin
- Greece (3):
  - Errikos Dunant Hospital Center-Fourth Department of Oncology and Clinical Trials Unit ( Site 1301), Athens, Attica
  - THORACIC GENERAL HOSPITAL OF ATHENS "I SOTIRIA"-3rd Dept of Internal Medicine and Laboratory, Oncol ( Site 1300), Athens, Attica
  - European Interbalkan Medical Center-Oncology Department ( Site 1302), Thessaloniki
- Hungary (5):
  - Pécsi Tudományegyetem Klinikai Központ-Onkoterápiás Intézet ( Site 1402), Pécs, Baranya
  - Bacs-Kiskun Varmegyei Oktatokorhaz-Onkoradiologiai Kozpont ( Site 1401), Kecskemét, Bács-Kiskun county
  - Gyor-Moson-Sopron Varmegyei Petz Aladar Egyetemi Oktato Korhaz - Pulmonologia Osztaly ( Site 1404), Győr, Győr-Moson-Sopron
  - Reformatus Pulmonologiai Centrum ( Site 1405), Törökbálint, Pest County
  - Somogy Varmegyei Kaposi Mor Oktato Korhaz -Onkologiai Kozpont ( Site 1407), Kaposvár, Somogy County
- Tallaght University Hospital ( Site 3903), Dublin, Ireland
- Italy (10):
  - Instituto Tumori Giovanni Paolo II-SSD Oncologia Medica per la Patologia Toracica ( Site 1507), Bari, Apulia
  - CRO-IRCCS-Clinical Oncology ( Site 1510), Aviano, Friuli Venezia Giulia
  - P.O. "S. Maria della Misericordia" Azienda Sanitaria Univers-Oncology Department ( Site 1506), Udine, Friuli Venezia Giulia
  - Fondazione IRCCS Istituto Nazionale dei Tumori-Struttura Complessa Oncologia Medica 1 ( Site 1504), Milan, Lombardy
  - ASST Grande Ospedale Metropolitano Niguarda-Oncologia Falck ( Site 1511), Milan, Milano
  - A.O.R.N. Ospedale dei Colli - Monaldi V.-U.O.C Pneumologia Oncologica DH PNL ONC ( Site 1508), Naples, Napoli
  - POLICLINICO "G. RODOLICO"-UOC Oncologia Medica ( Site 1503), Catania, Sicily
  - AO Santa Maria della Misericordia-Oncology Department ( Site 1501), Perugia, Umbria
  - Azienda Ospedaliera Santa Croce e Carle ( Site 1500), Cuneo
  - Azienda Ospedaliero Universitaria Maggiore della Carità ( Site 1502), Novara
- Japan (11):
  - Nagoya University Hospital ( Site 3810), Nagoya, Aichi-ken
  - Hirosaki University Hospital ( Site 3808), Hirosaki, Aomori
  - National Cancer Center Hospital East ( Site 3800), Kashiwa, Chiba
  - Hyogo Cancer Center ( Site 3809), Akashi, Hyōgo
  - St. Marianna University Hospital ( Site 3802), Kawasaki, Kanagawa
  - Kanagawa Cancer Center ( Site 3801), Yokohama, Kanagawa
  - Sendai Kousei Hospital ( Site 3805), Sendai, Miyagi
  - Kansai Medical University Hospital ( Site 3806), Hirakata, Osaka
  - Kindai University Hospital ( Site 3803), Sakai, Osaka
  - Hiroshima University Hospital ( Site 3804), Hiroshima
  - Okayama University Hospital ( Site 3807), Okayama
- RIGA EAST UNIVERSITY HOSPITAL ,Oncology Centre of Latvia ( Site 1600), Riga, Latvia
- Lithuania (2):
  - Hospital of Lithuanian University of Health Sciences Kauno klinikos-Pulmonology ( Site 1701), Kaunas, Kaunas County
  - Vilnius University Hospital Santaros Clinics Affiliate - National Cancer Center ( Site 1700), Vilnius
- Malaysia (5):
  - University Malaya Medical Centre ( Site 3502), Lembah Pantai, Kuala Lumpur
  - National Cancer Institute-Radiotherapy and Oncology ( Site 3506), Putrajaya, Kuala Lumpur
  - Hospital Tengku Ampuan Afzan ( Site 3504), Kuantan, Pahang
  - Hospital Pulau Pinang ( Site 3505), George Town, Pulau Pinang
  - Sarawak General Hospital ( Site 3500), Kuching, Sarawak
- Mexico (6):
  - CIO - Centro de Inmuno-Oncología de Occidente ( Site 3403), Guadalajara, Jalisco
  - Hospital Universitario "Dr. Jose Eleuterio Gonzalez"-Hematologia and Oncologia ( Site 3408), Monterrey, Nuevo León
  - Unidad de Mastologia Avanzada de Chihuahua S.A de C.V ( Site 3402), Chihuahua City
  - Mediadvance Clinical ( Site 3404), Chihuahua City
  - Oaxaca Site Management Organization S.C. ( Site 3407), Oaxaca City
  - Centro de Investigacion Clinica de Oaxaca ( Site 3401), Oaxaca City
- New Zealand (2):
  - New Zealand Clinical Research (Christchurch) ( Site 0300), Christchurch, Canterbury
  - Harbour Cancer & Wellness ( Site 0301), Auckland
- Norway (3):
  - Akershus Universitetssykehus-Avdeling for lungesykdommer ( Site 1900), Lørenskog, Akershus
  - Drammen Sykehus, Vestre Viken HF ( Site 1903), Drammen, Buskerud
  - Stavanger Universitetssykehus ( Site 1901), Stavanger, Rogaland
- Philippines (3):
  - Metro Davao Medical and Research Center ( Site 3602), Davao City, Davao Del Sur
  - ST. LUKE'S MEDICAL CENTER ( Site 3606), Quezon City, National Capital Region
  - CARDINAL SANTOS MEDICAL CENTER-Research Room ( Site 3601), San Juan City, Metro Manila, National Capital Region
- Poland (8):
  - Wielkopolskie Centrum Pulmonologii i Torakochirurgii-Oddzial Onkologii Klinicznej z Pododdzialem Dz ( Site 2002), Poznan, Greater Poland Voivodeship
  - Centrum Onkologii im. Prof. Franciszka Lukaszczyka-Ambulatorium Chemioterapii ( Site 2003), Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Krakowski Szpital Specjalistyczny im. Jana Pawła II-Oddział Kliniczny Chirurgii Klatki Piersiowej i ( Site 2011), Krakow, Lesser Poland Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - P-Klinika Nowotworow Pluca i Klatki Pier ( Site 2000), Warsaw, Masovian Voivodeship
  - Wojewodzki Szpital im. Sw. Ojca Pio w Przemyslu ( Site 2001), Przemyśl, Podkarpackie Voivodeship
  - Bialostockie Centrum Onkologii ( Site 2005), Bialystok, Podlaskie Voivodeship
  - Uniwersyteckie Centrum Kliniczne ( Site 2013), Gdansk, Pomeranian Voivodeship
  - Warmińsko - Mazurskie Centrum Chorób Płuc w Olsztynie-Oddzial Onkologii z Pododdzialem Chemioterapii ( Site 2008), Olsztyn, Warmian-Masurian Voivodeship
- Portugal (2):
  - Unidade Local de Saude de Santa Maria - Hospital Pulido Valente ( Site 2703), Lisbon, Lisbon District
  - Instituto Português de Oncologia do Porto Francisco Gentil, EPE ( Site 2702), Porto
- Slovakia (4):
  - Fakultna nemocnica s poliklinikou F.D.Roosevelta Banska Bystrica ( Site 2202), Banská Bystrica, Banská Bystrica Region
  - Univerzitná nemocnica Bratislava - Nemocnica Ružinov ( Site 2201), Bratislava, Bratislava Region
  - Nemocnica BORY a. s. ( Site 2205), Bratislava, Bratislava Region
  - Vychodoslovensky Onkologicky ustav a.s. ( Site 2200), Košice, Košice Region
- South Korea (8):
  - National Cancer Center-Lung Cancer Center ( Site 0403), Goyang-si, Kyonggi-do
  - Seoul National University Bundang Hospital-Medical Oncology ( Site 0404), Seongnam, Kyonggi-do
  - The Catholic University Of Korea St. Vincent's Hospital-Medical Oncology ( Site 0406), Suwon, Kyonggi-do
  - Chungbuk National University Hospital-Internal medicine ( Site 0402), Cheongju-si, North Chungcheong
  - Keimyung University Dongsan Hospital CRC room 1 ( Site 0407), Daegu, Taegu-Kwangyokshi
  - Seoul National University Hospital ( Site 0400), Seoul
  - Asan Medical Center-Department of Oncology ( Site 0405), Seoul
  - Samsung Medical Center ( Site 0401), Seoul
- Spain (6):
  - Institut Català d'Oncologia - L'Hospitalet-Medical Oncology ( Site 2401), L'Hospitalet de Llobregat, Barcelona
  - HOSPITAL UNIVERSITARIO QUIRONSALUD MADRID-ONCOLOGIA MEDICA ( Site 2402), Pozuelo de Alarcón, Madrid
  - HOSPITAL UNIVERSITARIO PUERTA DE HIERRO MAJADAHONDA-Medical Oncology ( Site 2403), Majadahonda, Madrid, Comunidad de
  - Hospital Quirón Málaga ( Site 2405), Málaga, Malaga
  - Hospital Universitari Vall d'Hebron-Departamento de Oncologia- VHIO ( Site 2400), Barcelona
  - Hospital Universitario Virgen Macarena-Unidad de Investigación Oncológica ( Site 2404), Seville
- Taiwan (7):
  - National Taiwan University Cancer Center (NTUCC) ( Site 0500), Taipei City, Taipei
  - Changhua Christian Hospital ( Site 0504), Changhua
  - National Taiwan University Hospital - Hsinchu branch ( Site 0501), Hsinchu
  - Taichung Veterans General Hospital-Chest ( Site 0503), Taichung
  - National Cheng Kung University Hospital-Clinical Trial Center ( Site 0505), Tainan
  - National Taiwan University Hospital-Oncology ( Site 0506), Taipei
  - Taipei Medical University Hospital ( Site 0502), Taipei
- Turkey (Türkiye) (7):
  - Medipol Mega Universite Hastanesi-oncology ( Site 2105), Stanbul, Istanbul
  - Ege Universitesi Hastanesi-Chest Diseases Department ( Site 2107), Bornova, İzmir
  - Hacettepe Universite Hastaneleri-oncology hospital ( Site 2100), Ankara
  - Memorial Ankara Hastanesi-Medical Oncology ( Site 2103), Ankara
  - Liv Hospital Ankara-Oncology ( Site 2104), Ankara
  - Ankara Bilkent Şehir Hastanesi-Medical Oncology ( Site 2101), Ankara
  - TC Saglik Bakanligi Goztepe Prof. Dr. Suleyman Yalcin Sehir Hastanesi-oncology ( Site 2102), Istanbul

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26311&tenant=MT_MSD_9011